CLINICAL TRIAL: NCT04241510
Title: Effects of Kinesio Taping Techniques on Pulmonary Parameters and Functional Exercise Capacity in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Kinesio Taping Techniques in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Burcu Camcıoğlu Yılmaz, PT, PhD, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KPR1
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Mechanical Correction; Facilitation; Thoracic Taping; Kinesio Taping; Respiratory Muscle Strength; Pulmonary Functions; Functional Exercise Capacity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Prospective, Double-Blinded, Randomized Crossover Study
Who Masked: Participant, Outcomes Assessor
Masking Description: Evaluation of patients after taping application will be done by another physiotherapist who does not know the taping techniques and also cannot see the taped area by clothes of patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Facilitation Tape (Active Comparator): Diaphragm and Intercostal muscles will be taped with facilitation technique. After 30 minutes of application patients will be evaulated for pulmonary parameters, functional exercise capacity and dyspnea.
  Interventions: Device: Kinesio Taping
- Mechanical Correction Tape (Active Comparator): Thorax will be taped with mechanical correction technique. After 30 minutes of application patients will be evaulated for pulmonary parameters, functional exercise capacity and dyspnea.
  Interventions: Device: Kinesio Taping
- No Tape (No Intervention): Patients will be evaulated for pulmonary parameters, functional exercise capacity and dyspnea with no tape.

INTERVENTIONS:
Device: Kinesio Taping — Kinesio Taping is a special taping method developed by Dr. Kenzo Kase in 1973. This technique triggers natural healing responses of human body by activating nervous and circulatory systems. The tapes are thin, latex-free, cotton, porous and anti-allergenic, with equal thickness of epidermis. It has elastic properites which allows the tape to elongate to %55-60 of its original lenght. Tape can be used up to 1 week even after sweating or cleaning with water. There are different application techniques for different purposes. Facilitation technique facilitates muscle contractions and supports muscle function. Mechancial correction technique is used for joint positioning and correcting motion of muscle-joint dynamics.
  Arms: Facilitation Tape; Mechanical Correction Tape

SUMMARY:
Study will investigate effects of two different kinesio taping techniques on pulmonary parameters of patients with COPD.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is an irreversible, progressive, treatable airway disease which causes dyspnea, wheezing, coughing and increased secretions in airways. Thoracic and respiratory mechanics are impaired, respiratory muscle strength and functional exercise capacity is decreased in patients with COPD. As a result dyspnea, limitation in activities of daily living, postural impairments, muscle length-strength relationship changes and increased mechanical loads on respiratory muscles occur. In literature it has been demonstrated that Kinesio Taping have therapeutic effects on respiratory functions and functional exercise capacity in patients with chronic neurological diseases who has additional respiratory impairments. Although there are several studies in literature investigating the effects of facilitation and inhibition taping techniques applied on respiratory muscles in patients with COPD, effects of thoracic and postural mechanical correction techniques as an alternative treatment modality in patients with COPD have not been investigated yet. In present study, effects of thoracic mechanical correction and facilitation taping techniques in patients with COPD will be investigated, and data will be collected for effects of thoracic mechanical correction taping on pulmonary parameters in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Male and female COPD patients aged between 40-80 years
* Diagnosed with COPD stage I-II-III-IV according to GOLD 2019 criterias
* Able to speak, understand and read Turkish language
* Volunteering to participate in study

Exclusion Criteria:

* Unstable or acutely exacerbated patients with COPD
* Alterations in medical treatment in last 6 months
* Having comorbidities that affect directly cardiopulmonary system, uncontrolled arterial hypertension, severe congestive heart failure, coronary arterial disease, heart valve disease
* Orthopaedic, neurological, psychiatric disease, peripheral/central nervous system diseases, mental retardation, antidepressants usage, metabolic impairments, malignancy
* Unable to cooperate for measurement and treatment techniques used in study
* Irritation, infection, allergic reaction, scarred burn or open wound around application area
* Enrolled in a comprehensive pulmonary rehabilitation program before study
* Application of Kinesio Tape to any body region in the past
* History of an open heart surgery or other thoracic surgeries

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Test | 30 minutes after every application
  Pulmonary functions will be evaulated in laboratory conditions. Dynamic lung volumes will be measured using standardized spirometric measurement regulations established by ATS/ERS guidelines.
Respiratory Muscle Strength | 30 minutes after every application
  Respiratory muscle strenght will be measured as Maximum Inspiratory Pressure & Maximum Expiratory Pressure with MicroMPM device. Measuring procedure will be held according to ERS guidelines. Measurements will be interpreted with Black and Hyatt's references.
Functional Exercise Capacity | 30 minutes after every application
  Functional exercise capacity will be measured with 6-minute walk test. Cardiovascular paremeters, dyspnea, respiratory rate and fatigue will be evaulated before, during and after the test .
Dyspnea | 30 minutes after each application
  Dyspnea in daily living was evaluated by the Modified Medical Research Council Dyspnea Scale. The scale consists in five statements that describe almost the entire range of dyspnea from none (Grade 0) to almost complete incapacity (Grade 4). Higher scores indicates increased dyspnea perception.

SECONDARY OUTCOMES:
Perception of Disease | 30 minutes after each application.
  COPD Assesment Test (CAT) will be used to evaulate patients perception of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Camcıoğlu Yılmaz, PT, PhD, Study Director — Muğla Sıtkı Koçman University; Metehan Sarıkaya, MSc. Student, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Muğla Sıtkı Koçman University Training and Research Hospital, Muğla, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Global Initiative for Chronic Obstructive Lung Disease (2019 Report). 2019;2-14
- [Background] Orozco-Levi M. Structure and function of the respiratory muscles in patients with COPD: impairment or adaptation? Eur Respir J Suppl. 2003 Nov;46:41s-51s. doi: 10.1183/09031936.03.00004607. PMID 14621106
- [Background] Kaneko H, Shiranita S, Horie J, Hayashi S. Reduced Chest and Abdominal Wall Mobility and Their Relationship to Lung Function, Respiratory Muscle Strength, and Exercise Tolerance in Subjects With COPD. Respir Care. 2016 Nov;61(11):1472-1480. doi: 10.4187/respcare.04742. Epub 2016 Oct 18. PMID 27794081
- [Background] Kenso Kase, Jim Wallis, Tsuyoshi Kase - Clinical Therapeutic Application Kinesio® Taping Manual. 2nd ed. Kinesio; 2003. 12-39 p.
- [Background] Kase K. Kenzo Kase. - Illustrated Kinesio Taping. In: 4th ed. p. 6-12, 72-5.
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Rostagno C, Gensini GF. Six minute walk test: a simple and useful test to evaluate functional capacity in patients with heart failure. Intern Emerg Med. 2008 Sep;3(3):205-12. doi: 10.1007/s11739-008-0130-6. Epub 2008 Feb 26. PMID 18299800
- [Background] Cheng SL, Lin CH, Wang CC, Chan MC, Hsu JY, Hang LW, Perng DW, Yu CJ, Wang HC; Taiwan Clinical Trial Consortium for Respiratory Disease (TCORE). Comparison between COPD Assessment Test (CAT) and modified Medical Research Council (mMRC) dyspnea scores for evaluation of clinical symptoms, comorbidities and medical resources utilization in COPD patients. J Formos Med Assoc. 2019 Jan;118(1 Pt 3):429-435. doi: 10.1016/j.jfma.2018.06.018. Epub 2018 Aug 25. PMID 30150099
- [Background] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Background] Yorgancioglu A, Polatli M, Aydemir O, Yilmaz Demirci N, Kirkil G, Nayci Atis S, Kokturk N, Uysal A, Akdemir SE, Ozgur ES, Gunakan G. [Reliability and validity of Turkish version of COPD assessment test]. Tuberk Toraks. 2012;60(4):314-20. doi: 10.5578/tt.4321. Turkish. PMID 23289460
- [Result] Kinesio Tape® Applied to the Thorax Augments Ventilatory Efficiency during Heavy Exercise. Int J Exerc Sci. 2013;6(2):8.
- [Result] Metin Okmen B, Sengoren Dikis O, Okmen K, Altan L, Yildiz T. Investigation of the effect of kinesiotaping on the respiratory function and depression in male patients with chronic obstructive pulmonary disease: a prospective, randomized, controlled, and single-blind study. Aging Male. 2020 Dec;23(5):648-654. doi: 10.1080/13685538.2019.1567703. Epub 2019 Feb 10. PMID 30739540
- [Result] Aydoğan Arslan S, Daşkapan AD, Özünlü Pekyavaş N, Sakızlı E. Effects of Kinesio Taping Applied to Diaphragm Muscle on Aerobic Exercise Capacity and Pulmonary Function in Sedentary Individuals. Anadolu Klin Tıp Bilim Derg. 2018;23(2):68-72.
- [Result] Zübeyir S, Nilüfer K, Burcu C, Onur A, Bahar K, Ufuk YS, et al. The Effect of Kinesiology Taping on Respiratory Muscle Strength. J Phys Ther Sci. 2012;24(3):241-4.
- [Result] Tomruk M, Keles E, Ozalevli S, Alpaydin AO. Effects of thoracic kinesio taping on pulmonary functions, respiratory muscle strength and functional capacity in patients with chronic obstructive pulmonary disease: A randomized controlled trial. Explore (NY). 2020 Sep-Oct;16(5):332-338. doi: 10.1016/j.explore.2019.08.018. Epub 2019 Sep 18. PMID 31611155
- [Result] Yoshida A, Kahanov L. The effect of kinesio taping on lower trunk range of motions. Res Sports Med. 2007 Apr-Jun;15(2):103-12. doi: 10.1080/15438620701405206. PMID 17578750
- [Result] Halseth T, McChesney JW, Debeliso M, Vaughn R, Lien J. The effects of kinesio taping on proprioception at the ankle. J Sports Sci Med. 2004 Mar 1;3(1):1-7. eCollection 2004 Mar. PMID 24497814
- [Result] Bostancı N., Yiğit Z., Baltacı G., Gürses H. Effects of kinesio taping method on pulmonary function, respiratory muscle strength and functional capacity in patients with chronic heart failure. Am J Respir Crit Care Med. 2018;197.
- [Result] Shih YF, Lee YF, Chen WY. Effects of Kinesiology Taping on Scapular Reposition Accuracy, Kinematics, and Muscle Activity in Athletes With Shoulder Impingement Syndrome: A Randomized Controlled Study. J Sport Rehabil. 2018 Nov 1;27(6):560-569. doi: 10.1123/jsr.2017-0043. Epub 2018 Oct 15. PMID 29364027
- [Result] Han JT, Lee JH, Yoon CH. The mechanical effect of kinesiology tape on rounded shoulder posture in seated male workers: a single-blinded randomized controlled pilot study. Physiother Theory Pract. 2015 Feb;31(2):120-5. doi: 10.3109/09593985.2014.960054. Epub 2014 Sep 29. PMID 25264014
- [Result] Cools AM, Witvrouw EE, Danneels LA, Cambier DC. Does taping influence electromyographic muscle activity in the scapular rotators in healthy shoulders? Man Ther. 2002 Aug;7(3):154-62. doi: 10.1054/math.2002.0464. PMID 12372312
- [Result] Wang JS, Cho KH, Park SJ. The immediate effect of diaphragm taping with breathing exercise on muscle tone and stiffness of respiratory muscles and SpO2 in stroke patient. J Phys Ther Sci. 2017 Jun;29(6):970-973. doi: 10.1589/jpts.29.970. Epub 2017 Jun 7. PMID 28626302